CLINICAL TRIAL: NCT05467176
Title: A Multi-Center, Prospective, Observational Study of Patients Being Treated With ORGOVYX
Acronym: OPTYX
Status: Active, not recruiting | Type: Observational
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MVT-601-058
Record Dates: First submitted 2022-06-15; First posted 2022-07-20 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: relugolix; ORGOVYX; prostate cancer; OPTYX
MeSH Terms: conditions — Prostatic Neoplasms | interventions — relugolix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with Prostate Cancer: Patients with prostate cancer who are initiating treatment or have initiated treatment with ORGOVYX (per label instructions) within 1 month prior to enrollment and who remain on treatment at the time of enrollment.
  Interventions: Drug: Relugolix

INTERVENTIONS:
Drug: Relugolix — Relugolix 120-mg tablet administered orally once daily following an oral loading dose of 360 mg (3 x 120-mg tablets) on Day 1
  Other Names: TAK-385; MVT-601; RVT-601; T-1331285; ORGOVYX

SUMMARY:
This is a multi-center, prospective, observational study of patients being treated with ORGOVYX. The goal of this study is to generate real-world evidence about the safety and effectiveness of ORGOVYX in patients with prostate cancer in routine clinical care and the clinical course during treatment with and following cessation of ORGOVYX.

DETAILED DESCRIPTION:
This prospective observational cohort study will be conducted in patients who are initiating treatment or have initiated treatment with ORGOVYX within the 1 month prior to the time of study enrollment and who remain on treatment at the time of enrollment. The decision to initiate treatment with ORGOVYX should be made prior to study enrollment. The study is designed to better understand the actual experience of patients with prostate cancer treated with ORGOVYX by collecting data on treatment patterns, adherence, and selective safety data. Additionally, a better understanding of the trajectory of patients with prostate cancer following cessation of ORGOVYX therapy will be gained by observing the clinical course of the disease, health outcomes, and health-related quality-of-life (HRQoL) in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with prostate cancer and initiating treatment with ORGOVYX at the time of enrollment or within 1 month prior to enrollment and who remain on treatment at enrollment
* Patients who are willing and able to complete PRO assessments during the study
* Patients who have reviewed and signed the informed consent form (ICF)

Exclusion Criteria:

* Patients with a history of surgical castration
* Patients with a medical or psychiatric condition that precludes participation in the opinion of the treating physician
* Patients whose original treatment plan is intended to be less than a total of 4 months of ORGOVYX

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prostate cancer who are initiating treatment or have initiated treatment with ORGOVYX within 1 month prior to enrollment and who remain on treatment at the time of enrollment
Sampling Method: Non-Probability Sample
Enrollment: 999 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Demographics | Up to 5 years
  Patient demographics
Selective Safety Data | Up to 5 years
  Incidence of treatment-related serious adverse events and any adverse events resulting in discontinuation of ORGOVYX as reported by physician or patient.
Health-Related Quality-of-Life Indicators | Up to 5 years
  Changes to health-related quality-of-life indicators as measured by patient-reported outcomes (PROs)
Clinical Characteristics | Up to 5 years
  Clinical characteristics of patients

SECONDARY OUTCOMES:
Clinical Course and Disease Progression | Up to 5 years
  Changes in disease stage and clinical treatment
Mortality | Up to 5 years
  Any deaths that occur during the study
Co-Morbidities | Up to 5 years
  Changes in co-morbidities (presence and/or severity) as assessed by patient's physician
Treatment Adherence | Up to 5 years
  Describe patient adherence and persistence including reasons for change with ORGOVYX treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sumitomo Pharma
Locations (96):
- United States (96):
  - Urology Centers of Alabama, Homewood, Alabama
  - Urology Associates of Mobile, Mobile, Alabama
  - Dignity Health, Phoenix, Arizona
  - Arizona Urology Specialists, PLLC, Tucson, Arizona
  - Arkansas Urology Research Center, Little Rock, Arkansas
  - City of Hope, Duarte, California
  - Urology Associates of Central California, Fresno, California
  - UCSD, La Jolla, California
  - USC Norris Cancer Center, Los Angeles, California
  - Tower Urology, Los Angeles, California
  - VA Greater Los Angeles Medical Center, Los Angeles, California
  - Tri Valley Urology, Murrieta, California
  - Genesis Research LLC, San Diego, California
  - Golden State Urology, Stockton, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - Banner MD Anderson Cancer Center, Greeley, Colorado
  - Colorado Urology, Lakewood, Colorado
  - Urology Associates, Lone Tree, Colorado
  - The Stamford Hospital, Stamford, Connecticut
  - Urologic Surgeons of Washington, Washington D.C., District of Columbia
  - MemorialCare, Long Beach Memorial Medical Center, Washington D.C., District of Columbia
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Manatee Medical Research Institute, LLC, Bradenton, Florida
  - Advanced Urology Institute, Daytona Beach, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - United Medical Group, Miami, Florida
  - SG Research LLC, Miami, Florida
  - Genesis Care USA, Naples, Florida
  - Florida Urology Partners, LLP, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Georgia Urology, Decatur, Georgia
  - PRiSMS Group LLC, Arlington Heights, Illinois
  - Associated Urological Specialists, Chicago Ridge, Illinois
  - Northwestern University, Evanston, Illinois
  - UroPartners Research, Glenview, Illinois
  - Comprehensive Urologic Care, Lake Barrington, Illinois
  - Duly Health and Care, Lisle, Illinois
  - Advanced Urology Associates, New Lenox, Illinois
  - Urology of Indiana, Carmel, Indiana
  - Urologic Specialists of Northwest Indiana, Merrillville, Indiana
  - Greater Regional Health, Creston, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Wichita Urology Group, P.A., Wichita, Kansas
  - Baptists Health Lexington, Lexington, Kentucky
  - Southern Urology, Lafayette, Louisiana
  - John Hopkins, Baltimore, Maryland
  - Chesapeake Urology Associates, Baltimore, Maryland
  - Maryland Oncology Hematology, Columbia, Maryland
  - Medstar Georgetown University Hospital, Columbia, Maryland
  - Michigan Institute of Urology, Troy, Michigan
  - GenesisCare USA, Troy, Michigan
  - Minnesota Urology, Woodbury, Minnesota
  - Specialty Clinical Research of St. Louis, St Louis, Missouri
  - Summit Medical Group, P.A. | New Jersey Urology, Berkeley Heights, New Jersey
  - AtlanticCare Cancer Institute, Egg Harbor, New Jersey
  - The Valley Hospital, Paramus, New Jersey
  - Regional Cancer Care Associates, Teaneck, New Jersey
  - Crystal Run Healthcare, Middletown, New York
  - Optum Medical Care, P. C., Mount Kisco, New York
  - Mount Sinai Hospital, New York, New York
  - SUNY Upstate Medical Institution, Syracuse, New York
  - Associated Medical Professionals of NY, PLLC, Syracuse, New York
  - Mohawk Valley Health Services, Utica, New York
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - Durham VA Healthcare, Durham, North Carolina
  - GenesisCare USA, Greenville, North Carolina
  - Associated Urologist of North Carolina, Raleigh, North Carolina
  - Clinical Inquest Center Ltd, Beavercreek, Ohio
  - NEO Urology Associates, Inc., Boardman, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals, Cleveland, Ohio
  - Central Ohio Urology Group, Gahanna, Ohio
  - Premier Clinical Research LLC dba STAT Research, Springboro, Ohio
  - The University of Toledo, Toledo, Ohio
  - Oregon Urology Institute, Springfield, Oregon
  - Spokenword Clinical Trials, Easton, Pennsylvania
  - Keystone Urology Specialist, Lancaster, Pennsylvania
  - GU, Inc., Latrobe, Pennsylvania
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - Lowcountry Urology Clinics, North Charleston, South Carolina
  - The Conrad Pearson Clinic, Germantown, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Urology Austin, Austin, Texas
  - Hmu, Crc Llc, Houston, Texas
  - MD Anderson, Houston, Texas
  - New Horizon Medical Group, LLC, Houston, Texas
  - Ascend Pharma Holdings, Houston, Texas
  - Urology San Antonio, P.A. dba USA Clinical Trials, San Antonio, Texas
  - The Urology Place, San Antonio, Texas
  - Potomac Urology Center, PC, Alexandria, Virginia
  - MedAtlantic, Richmond, Virginia
  - Urology of Virginia, PLLC, Virginia Beach, Virginia
  - Spokane Urology, P.S., Spokane, Washington
  - Wisconsin Institute of Urology, Neenah, Wisconsin
  - Aspirus, Wausau, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spratt DE, Dorff T, McKay RR, Lowentritt BH, Fallick M, Gatoulis SC, Flanders SC, Ross AE. Evaluating relugolix for the treatment of prostate cancer in real-world settings of care: the OPTYX study protocol. Future Oncol. 2024 Apr;20(12):727-738. doi: 10.2217/fon-2023-0748. Epub 2024 Mar 15. PMID 38488039